CLINICAL TRIAL: NCT00986271
Title: Extravascular Lung Water Index in Severe Sepsis
Acronym: EVLI in sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 97-0374B
Record Dates: First submitted 2009-09-27; First posted 2009-09-29 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2008-04

CONDITIONS: Severe Sepsis
Keywords: severe sepsis, intensive care units
MeSH Terms: conditions — Sepsis | interventions — Drug Delivery Systems

ARMS (1):
- With and without MODS developement (Other): EVLI was determinated by PiCCO plus system.
  Interventions: Procedure: EVLI was determinated by PiCCO plus system.

INTERVENTIONS:
Procedure: EVLI was determinated by PiCCO plus system.

SUMMARY:
To investigate whether extravascular lung water index (EVLI) is an independent predictor for multiorgan dysfunction syndrome (MODS) in patients with severe sepsis and to determine if increased EVLI may serve as an predictor for MODS and mortality in those patients.

ELIGIBILITY:
Inclusion Criteria:

* All enrolled patients were recruited consecutively on the day of MICU admission and within 24 hours of the diagnosis of severe sepsis.

Exclusion Criteria:

* Pregnancy,
* Age less than 18 years old, and
* Uncontrolled malignancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)

PRIMARY OUTCOMES:
Developement of MODS (multiorgan dysfunction syndrome) and mortality